CLINICAL TRIAL: NCT05273034
Title: Effect of the 1-hour Sepsis Bundle on In-hospital Mortality in Patients With Sepsis in the Emergency Department: a Randomized Controlled Trial
Brief Title: Effect of the 1-hour Sepsis Bundle on In-hospital Mortality in Patients With Sepsis in the Emergency Department
Acronym: 1BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APHP211023; IDRCB 2021-A01937-34 (Other: ANSM)
Record Dates: First submitted 2022-02-09; First posted 2022-03-10 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
Keywords: Sepsis; 1-hour sepsis bundle; Emergency department
MeSH Terms: conditions — Sepsis; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-h sepsis bundle (Experimental)
  Interventions: Procedure: 1-hour sepsis bundle
- Current practice (No Intervention)

INTERVENTIONS:
Procedure: 1-hour sepsis bundle — The sepsis management will be delivered in a timely manner within 60 minutes of ED triage including
  * usual test and treatment
  * blood culture
  * lactate measurement
  * broad spectrum antibiotics
  * In case of hypotension or lactate > 4, rapid administration of 30ml/kg crystalloid fluid resuscitation will be mandated
  * In case of initial elevated lactate (> 2 mmol/l), a second lactate measurement should be done after initial fluid resuscitation.
  Arms: 1-h sepsis bundle

SUMMARY:
Reducing the mortality and morbidity of sepsis is a worldwide priority for almost 20 years. Since an observational study in the NY state, which reported in-hospital mortality increased, associated with each supplemental hour to complete the sepsis bundle, SSC guidelines have decided in 2018 to recommend a short timeframe of 1-h to complete the sepsis bundle. This new recommendation is vividly debated due to a lack of evidences of its relevance. No trial has ever studied a sepsis intervention when applied as early as Emergency Department ED triage (newly recommended 1-h sepsis bundle consider time zero as time of ED triage).

The aim of this trial is to demonstrate that the early implementation at ED triage of the 1-hour bundle by ED physicians improves in-hospital mortality in patients with sepsis, and therefore provides the required robust evidence for the SSC guidance to enhance physicians and stakeholder adherence.

This is a superiority, international multicenter, open trial with a stepped wedge randomisation.

All centers will recruit adult emergency patients with suspicion of sepsis as defined by a suspicion of infection and suspicion of life threatening organ dysfunction (quick SOFA or SOFA ≥ 2, hypotension or hyperlactatemia).

According to the center period, the management of sepsis patients will be based either following the current recommended 1-hour sepsis bundle (intervention group) or at the discretion of the treating ED physician as in current routine practice (control group). There is no intervention that is "added" by the research.

DETAILED DESCRIPTION:
In Europe, one third of patients with sepsis and septic shock are admitted through the emergency department (ED), with an overall in-hospital mortality of 20%, and 90 days mortality of 25%. Reducing the mortality and morbidity of sepsis is thus a worldwide priority.

In 2016, the "Surviving Sepsis Campaign" (SSC), an international group of experts, recommended that physicians should complete the sepsis bundle in the first 3-h, which included blood culture, lactate measurement, broad spectrum antibiotics, and 30ml/kg fluid resuscitation in case of hypotension. Subsequently to the publication of a large retrospective study in NYC that reported a higher risk of mortality for each additional hour to complete the sepsis bundle, the 2018 update of the SSC guidelines moved further and recommended an even shorter timeframe of 1-h from ED triage to initiate the sepsis bundle. This new recommendation is vividly debated and several scientific societies, such as the SCCM, ACEP, and EUSEM have recommended that hospitals should not implement the one-hour sepsis bundle before having more evidence. Indeed, the quality of evidence supporting this new guidance was acknowledged overall as low to moderate and as requiring confirmatory studies. Moreover, no trial has ever studied a sepsis intervention when applied as early as ED triage (newly recommended 1-h sepsis bundle consider time zero as time of ED triage).

The primary objective of this trial is thus to demonstrate that the early implementation at ED triage of the 1-hour bundle by ED physicians improves in-hospital mortality in patients with sepsis, and therefore provides the required robust evidence for the SSC guidance to enhance physicians and stakeholder adherence. In-hospital mortality has been chosen as a primary endpoint in several major trials, such as ProCESS and ANDROMEDA SCHOCK. This in-hospital mortality will be truncated at 28 days because longer term to death may not reflect an effect of an early intervention. Furthermore, it has been described that mortality that occurs after hospital discharge may not be linked with the index acute disease, but rather mostly due to comorbidities (Frog ICU) and thus less relevant for assessing the efficacy of two early interventions.

Secondary objectives include the in-hospital morbidity, antibiotic exposure and fluid resuscitation, an all cause 28-day mortality with the implementation of the 1-hour sepsis bundle at ED triage vs practice in patients with sepsis in the ED.

The recommended 1-hour sepsis bundle (intervention group) carries the risk of over-exposition to antibiotics and excessive fluids resuscitation that may contribute to acute heart failure. However, the routine practice with longer time frame to complete the bundle carries the risk of sub-optimal treatment of sepsis with potential higher risk of mortality. Equipoise remains on which strategy carries the higher risk. Data from one large observational study suggest that each additional hour to the 1-hour sepsis bundle could increase mortality by an adjusted Odds Ratio of 1.04 (1.03 - 1.06).

This study will include patients that present to an ED with a suspicion of sepsis, as defined by the SEPSIS-3 consensus.

All centers will start in the control group for 4 weeks. Then, after every step of 4 weeks, two centers will switch to the intervention group, i.e. implementation at ED triage of the 1-h sepsis bundle. After the last center has switched for the intervention period, a last step of 4 weeks with all center in the intervention will be added. The order in which EDs will switch to the intervention will be randomized before the start of the trial.

The total duration of the study is planned to be 12 months (52 weeks) and 28 days with 24 centers expected.

Each participant with a suspicion of sepsis will be included and followed-up until hospital discharge at 28 days, whichever comes first. A follow-up at day 3 will be realised in order to collect components of the SOFA score and ICU status, and other secondary endpoints. If the patient is discharged before day 3, the last available hospital value will be used to calculate the SOFA score. The vital status of the patient will be assessed at day 28 or day of discharge alive.

Analysis will be performed at the end of the study after data review and before data base lock according to Intent to treat principle and with regard to cluster level randomisation.

ELIGIBILITY:
Inclusion Criteria:

* ED adult patients, with suspected infection
* Free given Oral consent given by the patient or by the trustworthy person / family member / close relative or inclusion in case of emergency.

AND at least one of the following:

* Serum lactate > 2.0 mmol/l
* Systolic blood pressure < 90 mmHg
* Suspicion of sepsis as defined by the SEPSIS-3 International consensus: life threatening organ dysfunction identified by a SOFA score of 2 at least or a quick SOFA score of 2 at least (altered consciousness, systolic blood pressure < 100 mmHg, respiratory rate > 22)
* For French sites, free given Oral consent given by the patient or by the trustworthy person / family member / close relative or inclusion in case of emergency. According to the Biomedical Research Law 14/2007 in Spain, the emergency consent is not apply. The written patient consent is mandatory.

Exclusion Criteria:

* Patient living in assisted-living home or nursing home or palliative center
* Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom
* Anticipated life expectancy < 3 months or "do not resuscitate" order
* Known acute heart failure
* No social security
* Pregnancy and breastfeeding
* Prisoners
* Participation in another interventional trial (RIPH 1 et 2)
* Patients that presented inclusion criteria more than 3 hours before inclusion
* Patient in whom antibiotics or fluid resuscitation has been started before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 873 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | truncated at day 28
  Safety Issue ? : Yes / No

SECONDARY OUTCOMES:
Amount of fluid resuscitation | in the first 24 hours
Acute heart failure | During the first 24 hours
  Acute heart failure defined by clinical signs of acute heart failure associated with either elevated brain natriuretic peptide or signs of pulmonary edema on chest imaging
SOFA score | Up to 3 days
  If the patient is discharged before day 3, the last available hospital value will be used to calculate the SOFA score.
ICU length of stay | Up to 3 days
Total number of days under mechanical ventilation, renal replacement therapy, and vasopressor-free | within 28 days
  Will be considered only during index hospitalisation
Undue antibiotic administration | Up to 3 days
  defined by introduction of antibiotic in the ED for patients in whom infectious disease was ruled out during hospital course
Mortality | at day 28
  death from all cause

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan FREUND, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided